CLINICAL TRIAL: NCT06119178
Title: EX-PRESS® P-50 and EX-PRESS® P-200
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: GLR516-P001
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EX-PRESS P-50: EX-PRESS P-50 filtration device implanted in one or both eyes during glaucoma surgery
  Interventions: Device: EX-PRESS P-50 filtration device
- EX-PRESS P-200: EX-PRESS P-200 filtration device implanted in one or both eyes during glaucoma surgery
  Interventions: Device: EX-PRESS P-200 filtration device

INTERVENTIONS:
Device: EX-PRESS P-50 filtration device — FDA-approved, stainless steel device with a 50-micron internal lumen size indicated for the reduction of intraocular pressure in glaucoma patients where medical and conventional surgical treatments have failed
  Groups: EX-PRESS P-50
Device: EX-PRESS P-200 filtration device — FDA-approved, stainless steel device with a 200-micron internal lumen size indicated for the reduction of intraocular pressure in glaucoma patients where medical and conventional surgical treatments have failed
  Groups: EX-PRESS P-200

SUMMARY:
The purpose of this Post-Market Clinical Follow-Up (PMCF) study is to assess long term clinical performance and safety outcomes for EX-PRESS Glaucoma Filtration Devices Models P-50 and P-200.

DETAILED DESCRIPTION:
This is a non-interventional/observational study designed as a retrospective chart review. Study sites will identify patient charts within their existing databases in a fair and consistent manner, e.g., reviewing all eligible charts in reverse chronological order by year of baseline visit. Patients meeting the eligibility criteria who have a minimum of 5 years of follow-up data since the implantation of the P-50 or P-200 device will be enrolled, including patients whose 5-year standard of care visit is scheduled during the study enrollment period.

The overall study duration is expected to be approximately 7 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an Institutional Review Board (IRB) / Independent Ethics Committee (IEC) approved informed consent form authorizing data collection prior to the review of any medical records;
* Implanted (one eye or both) with the EXPRESS P-50 or EXPRESS P-200 device per indications for use for at least 5 years;
* Have a minimum of 5 years of recorded follow-up data;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Enrolled in any clinical trial within the last 5 years;
* At the time of implantation:

  1. Presence of ocular disease such as uveitis, ocular infection, severe dry eye, severe blepharitis.
  2. Pre-existing ocular or systemic pathology that, in the opinion of the surgeon, is likely to cause postoperative complications following implantation of the device.
  3. Diagnosed with angle-closure glaucoma.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohorts will be selected from approximately 12 investigative sites located in the United States and/or outside the United States, approximately 4 countries.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Percentage reduction in intraocular pressure (IOP) from baseline | Baseline (preoperative), up to Year 5 postoperative
  IOP will be measured for each eye individually using applanation tonometry and recorded in millimeters mercury (mmHG).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (2):
- United States (2):
  - Boozman Hoff Regional Eye Clinic, Rogers, Arkansas
  - El Paso Eye Surgeons, PA, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No